CLINICAL TRIAL: NCT04342299
Title: The Antidepressant Advisor: A Decision Support System for UK Primary Care - a Feasibility Study: Study 3
Brief Title: The Antidepressant Advisor (Study 3): fMRI Study to Predict Treatment Response in Patients With Depression
Acronym: ADeSS_S3
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: NHS Lambeth Clinical Commissioning Group (Other)
Responsible Party: Principal Investigator, Dr Roland Zahn, Reader in the Neurocognitive Bases of Mood Disorders, Honorary Consultant Psychiatrist, King's College London
Other Study IDs: ADeSS_S3; PB-PG-0416-20039 (Other: National Institute for Health Research); 2064430 (Other: Medical Research Council); M816 (Other: Rosetrees Trust)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Antidepressant Medication; Treatment Resistance; Biomarker Candidates; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders: "Responders" are participants who show a reduction of depressive symptoms of at least 50%, as assessed by the self-rated Quick Inventory of Depressive Symptomatology (16-Item; self-report; QIDS-SR16) from baseline to follow-up.
  Please note that if the groups are skewed, a continuous measure (i.e. the difference between final and baseline depression scores) will be used rather than to categorise into responders and non-responders.
- Non-responders: "Non-responders" are participants who do not show a reduction of depressive symptoms of at least 50%, as assessed by the self-rated Quick Inventory of Depressive Symptomatology (16-Item; self-report; QIDS-SR16) from baseline to follow-up.
  Please note that if the groups are skewed, a continuous measure (i.e. the difference between final and baseline depression scores) will be used rather than to categorise into responders and non-responders.

SUMMARY:
This prospective observational study (ADeSS-Study3) investigates candidate biomarkers prospectively predicting response to antidepressant medications and prognosis in major depressive disorder (MDD). Currently, about half of MDD patients will not respond to the first course of selective serotonin reuptake inhibitors (SSRIs), while more than 40% will also not achieve remission after a second round of another SSRI. There are functional magnetic resonance imaging (fMRI) measures in several brain regions, showing clinical potential as predictors of response and non-response to SSRIs.

The overall aim of the study is to identify the neural signatures prospectively predicting poor prognosis in MDD patients after receiving four months of treatment in UK primary care. Specifically, it looks to evaluate four fMRI measures: 1) self-blame-selective subgenual cortex and ventral striatum connectivity with the right anterior temporal lobe; 2) pregenual anterior cingulate cortex activity in response to implicit emotional facial expressions; 3) amygdala activation in response to implicit emotional facial expressions; and 4) subgenual cingulate seed-based resting state.

In addition, a more specific objective of the study is to provide the proof-of-concept for using fMRI to prospectively predict which MDD patients will not benefit from SSRI antidepressant treatments in UK primary care. The long-term translational aim is to identify such patients and provide them with alternative treatments without delay by informing a decision support system with the information provided by these candidate biomarkers.

This study is linked to the Antidepressant Advisor Trial (ADeSS-Study 1: NCT03628027), in which the feasibility is evaluated of a novel computerised decision support system for antidepressant prescribing in MDD patients in a UK primary care setting.

DETAILED DESCRIPTION:
This prospective observational study focuses on identifying the neural signatures prospectively predicting poor prognosis in MDD patients after receiving four months of treatment in UK primary care.

It is expected that half of the patients will show a response to primary care treatment over the 16 weeks of the trial. This allows for comparison of baseline MRI scans of treatment responders with non-responders. The aim is to recruit at least n=12 in each group with complete data (responders vs non-responders), but if the groups are skewed, a continuous measure (i.e. the difference between final and baseline depression scores) will be used rather than to categorise into responders and non-responders. This sample size is considered sufficient for fMRI studies to run random-effect models. As there is no previous study from which effect sizes can be drawn, the study remains exploratory.

As this study aims to find candidate biomarkers predicting response to antidepressant treatment, it is important to define "response" and "antidepressant treatment". Response to treatment will be defined as a reduction of depressive symptom levels of at least 50%, as assessed by the self-rated Quick Inventory of Depressive Symptomatology (Self-report; 16-Item) from baseline to follow-up.

Due to the range of different antidepressants used in the main trial (Study 1), the primary analysis is to compare responders versus non-responders irrespective of treatment received which ensures the results are of pragmatic relevance to primary care treatment (considered as a complex multifaceted intervention for this study). The following antidepressants are likely to be prescribed in the study, either recommended by the algorithm or as initiated by general practitioners (GPs) without computerised decision support tool advice: sertraline (≥50mg; SSRI), escitalopram (≥10mg; SSRI), mirtazapine (≥30mg; alpha 2 antagonist; NaSSA; dual serotonin and norepinephrine agent), vortioxetine (≥10mg; multimodal), citalopram (≥20mg; SSRI), fluoxetine (≥20mg; SSRI), paroxetine (≥20mg; SSRI), venlafaxine (≥75mg; SSRI up to 150 mg and SNRI>150 mg), duloxetine (60mg; SNRI), therapeutic doses of tricyclics, and therapeutic doses of monoamine oxidase inhibitors.

Further analysis will be aimed at comparing response to another SSRI versus no response to another SSRI. Here, treatment with an SSRI will be defined as treatment with any of the earlier listed SSRIs, as well as low dose venlafaxine (up to 150mg). This includes individuals who started and subsequently stopped their SSRI or did not go up to an effective dose because of presumable side effects (intention-to-treat analysis). However, it excludes individuals whose SSRI has not been changed or whose SSRI dose has not been increased for the study period; individuals whose SSRI remained the same, but the dose increased are included. Individuals who were incompliant with their prescribed SSRI medication are included as their incompliance might be related to experiencing a poor benefit/side effect ratio (intention-to-treat analysis). Individuals who had medications with additional non-SSRI properties are excluded from this analysis (venlafaxine > 150 mg, mirtazapine > 15 mg, antipsychotics, lithium, tricyclics in therapeutic dose, monoamine oxidase inhibitors in therapeutic dose, or vortioxetine).

In order to investigate the general research aim, i.e. identifying the neural signatures prospectively predicting poor prognosis in MDD patients after receiving four months of treatment in UK primary care, the following specific neuroanatomical hypotheses are tested:

i) Moral sentiment task:

Following Lythe et al 2015, a longer version of this task predicted subsequent recurrence risk in remitted MDD patients. The authors found that patients with recurring MDD exhibited increased right superior anterior temporal cortex (RSATL) connectivity with the subgenual cortex (BA25), compared with MDD patients who remained in stable remission and a control group. In addition, the authors noted that RSATL hyper-connectivity with ventral putamen/claustrum, and the temporoparietal junction was distinctive of recurring MDD compared with stable MDD. The RSATL - temporoparietal junction hyper-connectivity did not survive a more stringent unpublished analysis applying a cluster-forming threshold of p=0.001 uncorrected as is now recommended.

Based on the inclusion criteria, it is expected that most patients in the current study will have recurring MDD. It is important to note that the study by Lythe et al 2015 was carried out in people with full remission. This suggests that their study may have been biased towards patients with an overall good prognosis for remission, as they will have responded to treatment before, and against patients with a chronic course of MDD. So, even though BA25 - ATL hyper-connectivity is associated with recurrence risk, it might also represent a marker of good prognosis for symptom remission.

Additional unpublished data collected by the Lythe et al 2015 authors was used to explore characteristics between those whose remission was attributable to serotonergic medications (n=36) and those who achieved remission through other means (n=28, e.g. psychotherapy or spontaneous remission), which was determined by the PI based on their recorded treatment history and blinded to the imaging results. Interestingly, people with a history of achieving remission using alternatives to serotonergic medications showed stronger hyper-connectivity of the right ventral striatum - RSATL compared to the others. In contrast, there was no difference between the two groups with regard to subgenual frontal - RSATL connectivity for self- versus other-blame. Notably, the groups were well-matched on demographic and clinical variables, which suggests that the lower ventral striatum - RSATL connectivity cannot be explained by other confounders and potentially is a genuine marker for serotonergic responders.

The Structured Clinical Interview for DSM-5 allows for the subtyping of MDD patients into subtypes: with anxious distress, with melancholic features (its operationalisation will be modified by requiring a lack of mood reactivity as a necessary criterion), and with atypical features. It is plausible that the prognosis varies for these MDD subtypes based on differences with regard to which part of the self-blaming bias-related neural network is more relevant. For example, MDD patients with anxious distress have been shown to have more anger towards others (captured as moderate and severe levels on the AMDP psychopathology interview) and benefit less from self-blame-related subgenual (BA25) - ATL-connectivity-reducing neurofeedback. Therefore, it is predicted that patients with anxious MDD are less likely to display self-blame-selective subgenual (BA25) - ATL hyper-connectivity.

Similarly, people with attention deficit hyperactivity disorder (ADHD), whose condition involves emotional instability which is captured as "affective lability" (moderate or severe levels) on the AMDP psychopathology interview, are predicted to show a lower likelihood of response to standard treatment in primary care with serotonergic antidepressants. It is predicted that they are more likely to experience anger towards others (captured as moderate and severe levels on the AMDP) and are therefore less likely to show self-blame-selective subgenual (BA25) - ATL hyper-connectivity.

Therefore, the following is hypothesised:

1. a) Self-blame-selective BA25 (using the Lythe et al 2015 results as a cluster-based ROI) - ATL hyper-connectivity (using the same right superior ATL seed as in Lythe et al 2015) will be associated with better prognosis after receiving four months of primary care treatment.

   b) Moreover, a lack of self-blame-selective hyper-connectivity will be associated with patients with anxious distress, who have a poorer prognosis and are more frequently encountered in treatment-resistant and chronic MDD samples. This type of sample is expected to be recruited for this study, whereas they are less likely to be recruited in remitted MDD studies such as the one published by Lythe et al 2015.
2. Self-blame-selective ventral striatum - ATL hyper-connectivity will be associated with poorer prognosis after receiving four months of primary care treatment. This is based on the fact that primary care mostly relies on SSRIs and SSRI response, which was retrospectively associated with a lack of self-blame-selective ventral striatum-ATL hyper-connectivity.
3. Lower self-blame-selective ventral striatum - ATL connectivity will be associated with better response to serotonergic medications. This is based on the comparison of those whose remission was attributable to serotonergic medications and those who achieved remission through other means (unpublished secondary data analysis of Lythe et al 2015 data).

ii) Implicit facial emotions task:

A) Following Godlewska et al 2018, the study team will probe the reproducibility of their findings regarding pregenual anterior cingulate cortex (pgACC) activity in response to implicit facial emotions as a predictor of response to treatment (six-weeks of treatment with escitalopram). The authors showed increased activity in the pgACC to sad versus happy faces in responders compared to non-responders.

Therefore, the hypothesis is that decreased activity in the pgACC ROI (obtained from the authors) to implicit sad versus happy faces is prospectively associated with poor prognosis after receiving four months of treatment.

B) In addition, this task allows to investigate amygdala activation as a potential predictor of response to treatment. Williams et al 2015 reported that responders to antidepressants (escitalopram (mean = 11.3 mg, sd = 6.7 mg), sertraline (mean = 59.3 mg, sd = 27.0 mg) and venlafaxine (mean = 92.3, sd = 32.2)) showed lower activation of the bilateral amygdala (Automated Anatomical Labelling (AAL) atlas ROI) for happy and left amygdala for sad faces compared to non-responders at baseline. Moreover, response to SSRIs was associated with lower activation of the amygdala for sad faces, and non-responders to venlafaxine displayed higher activation for sad faces. This finding is corroborated by a meta-analysis of functional predictors of treatment response, which linked increased activation in the right amygdala to an increased likelihood of poor response.

Therefore, the hypothesis is that increased activation of the amygdala for implicit sad and happy faces prospectively predicts poor prognosis after receiving four months of treatment, and the study team predicts that this increased amygdala response is more pronounced in patients with anxious distress given the link between increased arousal and anxiety, as well as significance and arousal signals being linked to amygdala activation in response to visual stimuli.

iii) Resting state fMRI:

Following Dunlop et al 2017, the study team will probe the reproducibility of their findings regarding subgenual cingulate cortex (SCC) connectivity as a predictor of response to treatment. The authors identified resting state functional connectivity between the SCC and three regions as a potential predictor: the left dorsal midbrain, the ventrolateral prefrontal cortex (VLPFC, Brodmann Area (BA) 47) and the left ventromedial frontopolar cortex (VMPFC, BA10). Absent and/or negative functional connectivity with the SCC was associated with remission following SSRI/SNRI treatment, whereas positive functional connectivity with the SCC was linked with treatment failure.

Therefore, the hypothesis is that positive functional connectivity between the SCC seed used by Dunlop - and the three ROIs to be obtained from the authors: VLPFC, SCC - VMPFC and SCC - dorsal midbrain prospectively predict poor prognosis after receiving four months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years +
* at least moderately severe major depressive syndrome on PHQ-9 (score 15 +)
* no plans to change GP practice
* able to complete self-report scales orally or in writing
* no previous prescription of mirtazapine or vortioxetine
* early treatment resistance as defined by 1) current or recent prescription (in the last 2 months) of any of the following antidepressants: citalopram, fluoxetine, sertraline, escitalopram, paroxetine, venlafaxine, or duloxetine AND 2) previous prescription of at least one other antidepressant out of the same list.

Exclusion Criteria:

* inability to consent to study
* unstable medical condition
* currently receiving specialist psychiatric treatment
* high suicide risk (MINI suicidality screen)
* past diagnosis of schizophrenia or schizo-affective disorder
* current psychotic symptoms (3 clinical screening questions)
* bipolar disorder
* currently at risk of being violent
* drug (modified PHQ) or alcohol abuse (PHQ) over last 6 months
* suspected central neurological condition
* pregnancy or insufficient contraception in women of childbearing age
* breastfeeding or within 6 months of giving birth in women of childbearing age
* both escitalopram and sertraline have already been prescribed
* MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Most participants will be recruited through GP practices, based in South London, taking part in the Antidepressant Advisor Trial (Study 1: NCT03628027).
  In addition, other participants will be recruited through online advertising. While it is essential for the larger clinical trial to recruit participants directly linked to a GP practice (to allow for comparison), this is not a requirement for this study.
  Control participants (no personal or family history of MDD) are recruited by asking enrolled participants to ask their partner or friend whether they would be interested. Using this approach, control participants are likely to be from the same socio-economic and educational backgrounds to the participants.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Baseline functional connectivity of the right superior anterior temporal lobe (RSATL) during self- vs. other-blame | 4 months
  Functional connectivity will be measured using an optimised and shortened version of the so-called moral sentiment task. Statistical Parametric Mapping 12 (SPM12) will be used to determine psychophysiological interactions between previously reported RSATL seed and previously identified clusters of connectivity in BA25 and putamen/claustrum. These two connectivity measures will be compared for self-blame vs. other-blame and entered as two predictor variables into a logistic regression model.
  The logistic regression model will include responder/non-responder as a binary outcome variable. Response to treatment will be defined as a reduction of depressive symptom levels of at least 50%, as assessed by the self-rated QIDS-SR16 from baseline to last follow-up.

SECONDARY OUTCOMES:
Baseline functional connectivity of the subgenual cingulate cortex (SCC) during resting state fMRI | 4 months
  Functional connectivity maps will be computed using the images for each participant by correlating average time course within the a priori subgenual frontal seed region with the time course in three a priori ROIs, as obtained from the Dunlop et al 2017 authors.
Baseline pregenual anterior cingulate cortex (pgACC) activity in response to implicit facial emotions | 4 months
  For this secondary outcome, the main ROI is the pgACC, as obtained from Godlewska et al 2018 authors.
  The task contrast of interest is the relative activation of sad vs happy faces. A 2-level analysis will be used to test the degree to which the change in neural activity in this contrast predicts response to treatment.
  The first level consists of sad vs happy contrast maps, calculated for each depressed subject. Second-level random effects analysis will assess whether this change in neural activity differs between responders and non-responders.
Baseline amygdala activation in response to implicit facial emotions | 4 months
  For this secondary outcome, the main ROI is the left and right amygdala, as defined by Automated Anatomical Labelling (AAL) atlas.
  SPM12 will be used to model the blood oxygen level-dependent (BOLD) effect for sad and happy blocks. In the first-level fixed-effect analysis, images will be derived for the contrast of sad vs neutral, and happy vs neutral. Individual contrast images will be normalised to standard space, which then will be used for second-level random effect analyses.
  Each participant's parameter estimates (beta weights) of amygdala activation will be extracted from the voxels that defined the cluster of significant activation. These represent an index of BOLD signal change for sad minus neutral, and happy minus neutral.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, IoPPN, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Harbi KS. Treatment-resistant depression: therapeutic trends, challenges, and future directions. Patient Prefer Adherence. 2012;6:369-88. doi: 10.2147/PPA.S29716. Epub 2012 May 1. PMID 22654508
- [Background] Dunlop BW, Rajendra JK, Craighead WE, Kelley ME, McGrath CL, Choi KS, Kinkead B, Nemeroff CB, Mayberg HS. Functional Connectivity of the Subcallosal Cingulate Cortex And Differential Outcomes to Treatment With Cognitive-Behavioral Therapy or Antidepressant Medication for Major Depressive Disorder. Am J Psychiatry. 2017 Jun 1;174(6):533-545. doi: 10.1176/appi.ajp.2016.16050518. Epub 2017 Mar 24. PMID 28335622
- [Background] Godlewska BR, Browning M, Norbury R, Igoumenou A, Cowen PJ, Harmer CJ. Predicting Treatment Response in Depression: The Role of Anterior Cingulate Cortex. Int J Neuropsychopharmacol. 2018 Nov 1;21(11):988-996. doi: 10.1093/ijnp/pyy069. PMID 30124867
- [Background] Williams LM, Korgaonkar MS, Song YC, Paton R, Eagles S, Goldstein-Piekarski A, Grieve SM, Harris AW, Usherwood T, Etkin A. Amygdala Reactivity to Emotional Faces in the Prediction of General and Medication-Specific Responses to Antidepressant Treatment in the Randomized iSPOT-D Trial. Neuropsychopharmacology. 2015 Sep;40(10):2398-408. doi: 10.1038/npp.2015.89. Epub 2015 Mar 31. PMID 25824424
- [Background] Lythe KE, Moll J, Gethin JA, Workman CI, Green S, Lambon Ralph MA, Deakin JF, Zahn R. Self-blame-Selective Hyperconnectivity Between Anterior Temporal and Subgenual Cortices and Prediction of Recurrent Depressive Episodes. JAMA Psychiatry. 2015 Nov;72(11):1119-26. doi: 10.1001/jamapsychiatry.2015.1813. PMID 26445229
- [Background] Flandin G, Friston KJ. Analysis of family-wise error rates in statistical parametric mapping using random field theory. Hum Brain Mapp. 2019 May;40(7):2052-2054. doi: 10.1002/hbm.23839. Epub 2017 Nov 1. PMID 29091338
- [Background] Thirion B, Pinel P, Meriaux S, Roche A, Dehaene S, Poline JB. Analysis of a large fMRI cohort: Statistical and methodological issues for group analyses. Neuroimage. 2007 Mar;35(1):105-20. doi: 10.1016/j.neuroimage.2006.11.054. Epub 2007 Jan 18. PMID 17239619
- [Background] Fu CH, Steiner H, Costafreda SG. Predictive neural biomarkers of clinical response in depression: a meta-analysis of functional and structural neuroimaging studies of pharmacological and psychological therapies. Neurobiol Dis. 2013 Apr;52:75-83. doi: 10.1016/j.nbd.2012.05.008. Epub 2012 Jun 1. PMID 22659303
- [Background] Pessoa L, Adolphs R. Emotion processing and the amygdala: from a 'low road' to 'many roads' of evaluating biological significance. Nat Rev Neurosci. 2010 Nov;11(11):773-83. doi: 10.1038/nrn2920. PMID 20959860